CLINICAL TRIAL: NCT03738709
Title: Occupational Therapy Group Program on Falls Prevention and Patient Education for the Older Adults Hospitalized in Service de Soins de Suite et de Réadaptation Gériatrique (SSRG) at Hôpitaux Universitaires de Strasbourg (HUS)
Brief Title: Occupational Therapy Group Program on Falls Prevention and Patient Education for the Older Adults Hospitalized
Acronym: ENCRAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 6790
Record Dates: First submitted 2018-10-26; First posted 2018-11-13 (Actual); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Fall
Keywords: Prevention; Group; Technical assistance; Fall; Occupational therapy; Hospitalization discharge
MeSH Terms: interventions — Occupational Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Occupational therapy group sessions (Experimental): In the collective experimental group, the care includes 6 group sessions of one hour each, programmed over 2 weeks and progressive courses.
  Interventions: Behavioral: Falls prevention and education giving a demonstration of the usage of technical assistance.
- Individual Occupational therapy sessions (Active Comparator): In the individual control group, care consists of 6 individual sessions of 45 minutes each, not programmed over 2 weeks and progressive courses.
  Interventions: Behavioral: Falls prevention and education giving a demonstration of the usage of technical assistance.

INTERVENTIONS:
Behavioral: Falls prevention and education giving a demonstration of the usage of technical assistance. — * Ecological trail to work on balance and walking.
  * Technical assistance presentation and try-outs within the therapeutic apartment.
  * Discussion on the perceived feelings over the exercises and the technical assistance submitted.
  * Falls Education and prevention, screening of the dangerous activities and education on the safe behaviours.
  Other Names: Occupational Therapy

SUMMARY:
The primary outcome is to assess the impact of the group program on falls prevention and patient education on home modifications and the implementation of technical assistance.

This study aims to demonstrate that a group program on falls prevention and patient education will improve the acceptance and the implementation of recommendations on technical assistance and home modifications following discharge after an hospitalization for fall.

The secondary outcome will measure the impact of the group program on the incidence of falls, the number of readmissions, fear of another fall and improvement in walking and balance skills.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female over 70 years old living at home and not in a nursing home, hospitalized after a fall or for a falls evaluation.
* Mini mental state examination score over or even 20/30.
* The person is planning to return home after discharge.

Exclusion Criteria:

* Decompensated medical pathologies.
* Severe chronical diseases with symptoms that are not stabilized by medical or non-medical treatments.
* Dizziness/vertigo linked to a vestibular or cerebellar disorder.
* Sensory disability preventing communication and participation in the group.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2018-12-04 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Number of technical assistance and home modifications implemented following discharge in both groups, in regard to the number of recommendations given during the hospitalization. | 1 month after hospitalization discharge (patient call #1)

SECONDARY OUTCOMES:
Number of technical assistance and home modifications implemented following discharge in both groups, in regard to the number of recommendations given during the hospitalization. | 6 months after hospitalization discharge (patient call #2)
Number of falls followed or not by an hospitalization since the discharge. | 6 months after the hospitalization discharge (patient call #2)
  The number of potential falls in the 6 months after discharge will be measured by a telephone call to the patient (if impossible, the call will be placed to his caregiver or nurse).
Fear of falling rate | At inclusion visit (visit 0; before the occupational therapy) and after the occupational therapy (visit 1; 2 weeks later)
  Fear of falling will be measured by the Falls Efficacy Scale I [FES-I] (score from 16 to 64; higher values represent a stronger fear of falling)
Evaluation of balance skills in daily living activities | At inclusion visit (visit 0; before the occupational therapy) and after the occupational therapy (visit 1; 2 weeks later)
  Balance skills will be measured by the "Equilibre et Vie Quotidienne" scale: scored from 6 (no danger) to 24 (high risk of fall with impossibility to realize the activities)
Evaluation of the walking by the "Stop Walking when Talking" test | At inclusion visit (visit 0; before the occupational therapy) and after the occupational therapy (visit 1; 2 weeks later)
  Positive test (pathological) if the subject stops walking when the therapist introduces a conversation
Evaluation of the motor skills by the Minimum Motor Test | At inclusion visit (visit 0; before the occupational therapy) and after the occupational therapy (visit 1; 2 weeks later)
  20 items distributed in 4 themes: mobility in decubitus, sitting position, standing position, walking.
  Each item rated from 0 (motor skill abnormal) to 1 (motor skill preserved) Total score from 0 to 20; higher values represent preserved motor skills
Evaluation of the walking speed by the Timed Up and Go test. | At inclusion visit (visit 0; before the occupational therapy) and after the occupational therapy (visit 1; 2 weeks later)
  The time of the course (in seconds) is retained as the final score. The test is positive if the score is 14 seconds or more, representing a risk of falling.
Evaluation of the number of footsteps in a 10 meters walk, by the Walk test on 10 meters. | At inclusion visit (visit 0; before the occupational therapy) and after the occupational therapy (visit 1; 2 weeks later)
  The score corresponds to the number of footsteps performed by the subject. Pathological score from 13 footsteps.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphanie BETTINELLI, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Soins de Suite et de Réadaptation Gériatrique - Ergothérapie -Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No